CLINICAL TRIAL: NCT03123653
Title: To Study the Efficacy of PEG-IFN Alpha in HBeAg Negative Chronic Hepatitis B Patients After Stopping Nucleotide Analogue Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HBV-01
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peg IFN 2b (Experimental): Peg IFN 2b 1.5mcg/kg once every week for 48 weeks.
  Interventions: Drug: Peg IFN 2b

INTERVENTIONS:
Drug: Peg IFN 2b — Peg IFN 2b 1.5mcg/kg once every week for 48 weeks

SUMMARY:
* Study population:Person with HBeAg negative CHB on TDF/ETV for more than 1 year
* Study design:Prospective,Interventional (single arm study)
* Sample size: All the patients fulfilling the inclusion criteria will be included in first 6 months and subsequently followed up for 2 years
* Intervention: Peg IFN 2b 1.5mcg/kg once every week for 48 weeks
* Monitoring and assessment: LFT,HBV DNA and HbsAg at baseline, 4 weeks, 12 weeks,24 weeks,48 weeks ,72 weeks and 96 weeks, CBC every month and Thyroid function Test every 3rd month
* Adverse effects: The most frequently reported side effects of IFN-based therapy are flu-like symptoms, headache, fatigue, myalgia, alopecia, and local reaction at the injection site. Peg-IFN have myelosuppressive effects; however, neutropenia\1000/mm3 and thrombocytopenia \500,000/ mm3 are not common unless patients already have cirrhosis

ELIGIBILITY:
Inclusion Criteria:

- HBeAg negative Chronic HBV infection who are having HBV DNA-undetectable. ALT <40 IU/ml No Advanced fibrosis[LSM <14 KPa] TDF/ETV >1 year Clinical Relapse after stopping NA will be defined as HBV DNA>2000IU/ml and ALT > 80IU

Exclusion Criteria:

- HBeAg+ CHB Pregnancy Cirrhosis on biopsy or LSM >14 Co-infection- HIV/HCV/HDV Immunosuppressive therapy Renal failure S.Bilirubin>2mg/dl Patient having neutropenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2020-09-17 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response-HBV DNA<2000IU/ml after stopping PEG IFN alpha | 6 months

SECONDARY OUTCOMES:
Loss of HBsAg after 48 weeks of PEG IFN alpha | 48 weeks
End treatment Response: HBV-DNA -undetectable after 48 weeks of PEG-IFN | 48 weeks
Sustained Off treatment Virological response defined as No clinical relapse during 1 year follow up after stopping therapy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No